CLINICAL TRIAL: NCT02602548
Title: The Incidence and Incubation Period of False Positive Cultures in Shoulder Surgery Study Protocol: A Pilot Study
Brief Title: The Incidence and Incubation Period of False Positive Cultures in Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Forte Sports Medicine and Orthopedics (Other)
Responsible Party: Principal Investigator, Gary Misamore, Orthopedic Surgeon, Forte Sports Medicine and Orthopedics
Other Study IDs: 1407463823
Record Dates: First submitted 2015-04-25; First posted 2015-11-11 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Infection
Keywords: Propionibacterium acnes; shoulder surgery; infection
MeSH Terms: conditions — Infections | interventions — Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open Shoulder Surgery: Culture
  Interventions: Other: Culture
- Arthroscopic Shoulder Surgery: Culture
  Interventions: Other: Culture

INTERVENTIONS:
Other: Culture — Specimens will be obtained and sent to the lab for cultures.

SUMMARY:
This study will describe the time point at which a positive culture from a patient who has undergone shoulder surgery should be treated as an infection versus a false positive result that should be disregarded. Intraoperative biopsies will be taken and cultured from 50 subjects who have undergone an "open" surgical procedure and 50 from subjects undergoing an arthroscopic procedure.

DETAILED DESCRIPTION:
Postoperative infection is a significant complication that requires timely identification and treatment. Indolent infections, such as those involving Propionibacterium acnes (P. acnes), pose a diagnostic dilemma as they present differently than the acute symptoms typically associated with most postoperative bone and joint infections. The workup of these suspected infections is also somewhat difficult, as these colonies are slow growing, necessitating that cultures be kept for an extended period of time. Previous studies have shown that positive cultures are typically identified between 7 and 13 days. In a recent study of patients undergoing primary shoulder arthroplasty, 41.8% of patients were found to have P. acnes growth from their joint fluid at a mean of 7 days (range 5-9 days). All of these patients were then treated immediately with 4 weeks of dual oral antibiotic therapy1.

As the incubation of laboratory cultures increases, there is the potential concern of false positive growth. Timely identification is critical in order to avoid performing unnecessary treatments on patients in whom no infection is actually present.

The investigators will enroll patients undergoing primary shoulder surgery for a clearly identified mechanical dysfunction, in which there is no clinical suspicion for infection. Infection should not exist in this population, making it an appropriate clinical sample in which to study results that the investigators would consider to be false positives.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary open and arthroscopic shoulder surgery in which there is a clear diagnosis of a mechanical problem that is felt to be amenable to surgical intervention and there is no suspicion of infection. Examples include, but are not limited to: rotator cuff tear, labral tear, instability, impingement, and osteoarthritis.

Exclusion Criteria:

* Prior shoulder surgery
* Prior glenohumeral injection within the last 6 months
* Systemic or shoulder inflammatory disorder
* Any clinical, imaging, or laboratory findings that raise suspicion of infection
* Minors
* Erythrocyte sedimentation rate (ESR) >15 mm/hr for males less than 50 years old, >20 mm/hr for males greater than 50 years old and females less than 50 years old, and >30 mm/hr for females greater than 50 years old
* C reactive protein (CRP) >1 mg/d,
* Procalcitonin (PCT) >0.05 ng/ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mechanical problems associated with their shoulder who elect to undergo shoulder surgery
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Incidence of positive cultures | 28 days

SECONDARY OUTCOMES:
Incubation time clarification for culture growth if it occurs | Less than or equal to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary Misamore, MD, Principal Investigator — Forte Sports Medicine and Orthopedics

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Butler-Wu SM, Burns EM, Pottinger PS, Magaret AS, Rakeman JL, Matsen FA 3rd, Cookson BT. Optimization of periprosthetic culture for diagnosis of Propionibacterium acnes prosthetic joint infection. J Clin Microbiol. 2011 Jul;49(7):2490-5. doi: 10.1128/JCM.00450-11. Epub 2011 May 4. PMID 21543562
- [Background] Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. doi: 10.1016/j.jse.2012.07.007. Epub 2012 Sep 13. PMID 22981447